CLINICAL TRIAL: NCT01268306
Title: A Single-site, Open-Label Prospective Evaluation of Biocompatibility and Corneal Staining Associated With Use of Bausch & Lomb (B+L) BioTrue Contact Lens Multi-purpose Solution (MPS) and B+L PureVision Contact Lenses.
Brief Title: Study of the Presence and Extent of Corneal Disturbance Associated With B+L Biotrue MPS Used With B+L PureVision Lenses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Epstein, Arthur B., OD, FAAO (Individual)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CLC-01
Record Dates: First submitted 2010-12-28; First posted 2010-12-30 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Keratitis
Keywords: contact lens; corneal staining; fluorescein staining; preservatives; keratitis; punctate keratopathy; superficial punctate keratopathy; SPK
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- B+L Biotrue MPS and B+L PureVision (Experimental): Successful contact lens wearers switched to B&L BioTrue MPS while wearing B+L PureVision lenses
  Interventions: Device: B+L Biotrue MPS and B+L PureVision

INTERVENTIONS:
Device: B+L Biotrue MPS and B+L PureVision — Subjects use Bausch & Lomb (B+L) Biotrue MPS with B+L PureVision contact lenses
  Other Names: B+L Biotrue; B+L PureVision

SUMMARY:
Corneal epithelial disruption, commonly termed "corneal staining" has been frequently associated with contact lens wear. Previous research has demonstrated higher levels of observed corneal staining when certain combinations of contact lenses and lens care products are used, particularly under daily wear regimens. B+L lenses made from Balafilcon (PureVision) have been associated with the highest rates of observed staining. Additionally, polyhexamethylene biguanide (PHMB) based lens care products, specifically B+L ReNu MultiPlus have been implicated in higher rates of staining. In general, many lenses constructed from newer, silicone hydrogel (SiHy) materials appear more susceptible to increased rates and amounts of corneal staining.

Although the clinical significance of staining is debated, most clinicians agree that less staining is preferable to greater amounts of staining. Advances in understanding as well as the specifics of lens care product formulation ideally will have resulted in design of newer products that minimize corneal staining and maximize product performance. This study will examine rates of corneal staining using B+L's recently introduced lens care product: BioTrue with the B+L PureVision lens which has previously been associated with the highest levels of staining.

DETAILED DESCRIPTION:
Corneal epithelial disruption, commonly termed "corneal staining" has been frequently associated with contact lens wear. Previous research has demonstrated higher levels of observed corneal staining when certain combinations of contact lenses and lens care products are used, particularly under daily wear regimens. B+L lenses made from Balafilcon (PureVision) have been associated with the highest rates of observed staining. Additionally, polyhexamethylene biguanide (PHMB) based lens care products, specifically B+L ReNu MultiPlus have been implicated in higher rates of staining. In general, many lenses constructed from newer, silicone hydrogel (SiHy) materials appear more susceptible to increased rates and amounts of corneal staining.

Although the clinical significance of staining is debated, most clinicians agree that less staining is preferable to greater amounts of staining. Advances in understanding as well as the specifics of lens care product formulation ideally will have resulted in design of newer products that minimize corneal staining and maximize product performance. This study will examine rates of corneal staining using B+L's recently introduced lens care product: BioTrue with the B+L PureVision lens which has previously been associated with the highest levels of staining.

This pilot study is intended to assess the presence of corneal staining among patients who are using BioTrue solution

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent document must be read, signed and dated by the patient or legally authorized representative.
2. Subjects 18 years of age or older.
3. Subjects may be of either sex and of any race.
4. History (within the past 6 months) of successful soft contact lens wear.
5. Subjects must be free of any ocular disorder that would contraindicate contact lens wear
6. Subjects must have grade 1 (trace) or less corneal staining at baseline measurement as determined by the investigator or subinvestigator
7. Ocular health within normal limits as determined by the investigator or subinvestigator.
8. Willing to wear test contact lenses and use test lens care product throughout the length of the study period.

Exclusion Criteria:

1. Inability to be properly fitted with test lenses.
2. Inability to comfortably tolerate test lenses or lens care product.
3. Inability or unwillingness to follow all study instructions and complete study visits as required.
4. Greater than grade 1 (trace) staining in any quadrant at baseline examination.
5. Presumed or actual ocular infection (bacterial, viral, or fungal) or history of ocular herpes in either eye as determined by subject history and/or examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur B. Epstein, OD, Principal Investigator
Locations (1):
- Joel J. Ackerman, OD, PC, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects randomly recruited from contact lens wearing population in an optometric practice
Pre-assignment Details: Patients with spherical contact lens corrections who achieved acceptable acuity with test lenses were offered study participation.
Groups:
- Bausch & Lomb (B+L) Biotrue MPS With B+L PureVision Lenses: Use of B+L Biotrue multipurpose solution (MPS) with PureVision contact lenses : Subjects use Bausch & Lomb (B+L) Biotrue MPS with B+L PureVision contact lenses
Period: Overall Study
Arm/Group | Bausch & Lomb (B+L) Biotrue MPS With B+L PureVision Lenses
Started | 8
Completed | 7
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bausch & Lomb (B+L) Biotrue MPS With B+L PureVision Lenses
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Wiith Corneal Staining
Description: The number of participants who have disturbance of their corneal epithelium visualized by using applied sodium fluorescein solution (as a disclosing agent) evaluated by slit lamp biomicroscopy. Clinically significant staining is described as sufficiently diffuse and deep to pose potential risk of infection by the examiners assessment.
Time Frame: 2-4 hours after contact lens insertion
Population: Subjects who returned for examination post-challenge in the allotted time and who had observable corneal staining on slit lamp examination
Measure: Number; unit: participants
Arm/Group | Bausch & Lomb (B+L) Biotrue MPS With B+L PureVision Lenses
Number analyzed (Participants) | 7
participants
  Clinically signficant staining | 1
  Clinically insigificant staining | 6

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Bausch & Lomb (B+L) Biotrue MPS With B+L PureVision Lenses
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Pilot study with insignificant subject population for statistical analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No